CLINICAL TRIAL: NCT01933022
Title: An Exploratory, Open Label, Single-arm Study to Evaluate the Effect of Eligard® 6-month on Biomarkers of Disease in Patients With Metastatic Prostate Cancer
Brief Title: A Study in Patients With Metastatic Prostate Cancer to Assess How the Drug Eligard®, Affects Certain Markers in Blood and Urine, Which Are Indicators for the Disease
Acronym: EFFECT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Termination due to high current screen rate failure and unreliable PSA mRNA assay.
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EGD-EC-005; 2012-000101-69 (EudraCT Number)
Record Dates: First submitted 2013-08-28; First posted 2013-08-30 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Prostate Cancer
Keywords: Exploratory; Biomarkers; Eligard; Metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — luprolide acetate gel depot; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm: Eligard (Other): Single Arm
  Interventions: Drug: Eligard

INTERVENTIONS:
Drug: Eligard — Subcutaneous Injection
  Other Names: Leuprorelin acetate

SUMMARY:
The purpose of this study is to investigate the effect of the study medication (Eligard®) on cancer markers (in the blood) of prostate cancer.

DETAILED DESCRIPTION:
The main objective of the study is to explore the effect of Eligard® on the following prostate cancer biomarkers:

Testosterone in serum, Prostate Specific Antigen (PSA) in serum, Prostate Cancer Antigen (PCA3 score) in urine, PSA mRNA in blood/Peripheral Blood Mononuclear Cell (PBMC), PCA3 mRNA in blood/PBMC, Transmembrane protease, serine 2-Ets Related Gene (TMPRSS2-ERG) mRNA in blood/PBMC

A blood sample for RNA analysis will also be collected and stored for future investigation in patients giving specific informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed metastatic prostate cancer for whom androgen deprivation therapy (ADT) is indicated.
* Non-castrate level of testosterone (≥ 8 nmol/L (230 ng/dL)) at screening.
* Serum PSA ≥ 5 ng/mL at screening.
* Eastern Cooperative Oncology Group (ECOG) score of 0-2
* A life expectancy of at least 12 months.
* Is able to tolerate injection of study drug and comply with the study requirements.
* Positive blood PSA mRNA at screening. A positive PSA mRNA in PBMCs (defined as exceeding the Limit of Detection [LoD] for the central lab assay, i.e. ≥ 10 copies per Polymerase Chain Reaction, PCR).

Exclusion Criteria:

* History of bilateral orchidectomy.
* History of any hormonal treatment/therapy with GnRH agonist, GnRH anti-agonist within 6 months of enrolment.
* Treatment with anti-androgens (except where used to prevent testosterone flare up, starting up to 2 weeks prior to Eligard injection, according to local treatment guidelines), 5-α reductase inhibitors, estrogens and/or other any investigational hormone-derivative within 3 months of enrolment or 5-times the half-life, whichever is longer.
* Any previous treatment with chemotherapy treatment for prostate cancer prior to the screening visit or within 6 months prior to screening for any other cancer.
* Patients previously treated for cancer with hormonal therapy in whom treatment was stopped due to lack of efficacy, progression of the disease or lack of tolerability.
* Previous treatments for cancer (including prostate cancer) within 6 months prior to enrolment: immunotherapy, external beam radiotherapy, brachytherapy, thermotherapy, or biological response modifiers (e.g. cytokines).
* Known or suspected spinal cord compression or evidence of spinal metastases with risk of spinal compression.
* Uni- or bilateral ureteric obstruction.
* Requiring concomitant use of anti-androgens during the course of the study (except where used to prevent testosterone flare up, starting up to 2 weeks prior to Eligard injection and continuing for up to 3 weeks, according to local treatment guidelines).
* Previous or concomitant malignancies at other sites except effectively treated non-melanoma skin cancer or an effectively treated malignancy that has been in remission for at least 5 years.
* Major surgery within 2 months prior to enrolment.
* Total bilirubin > 1.5 times the upper limit of normal (ULN) at screening. This will not apply to subjects with Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of evidence of hemolysis or hepatic pathology), who will be allowed in consultation with the sponsor.
* Participation in any clinical study within ≤ 1 month prior to screening (or 5 half lives of the drugs under investigation, whichever is greater).
* Not available for follow-up assessments or unable to comply with study requirements.
* Known or suspected hypersensitivity to leuprorelin acetate, to other GnRH agonists or to any of the excipients of Eligard.
* Male subjects who are intending to donate sperm within 9 months following the injection of Eligard
* Male subjects and their female spouses/partners who are of childbearing potential and are NOT using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continuing for 9 months from the time of the Eligard injection. Acceptable forms include:

  * Established use of oral, injected or implanted hormonal methods of contraception.
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
  * Barrier methods of contraception: Condom OR Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
* Absolute neutrophil count < 1,500/μL, platelet count < 100,000/μL, and hemoglobin < 5.6 mmol/L (9 g/dL) at screening.
* Alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) > 2 times ULN at screening.
* Creatinine > 177 μmol/L (2 mg/dL) at screening.
* Albumin ≤ 30 g/L (3.0 g/dL) at screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of Testosterone levels in serum | Baseline to 6 months
Changes from baseline of PSA level in serum | Baseline to 6 months
Changes from baseline of PCA3 score in urine | Baseline to 6 months
Changes from baseline of Number of PSA mRNA copies in blood/PBMC | Baseline to 6 months
Changes from baseline of Number of PCA3 mRNA copies in blood/PBMC | Baseline to 6 months
Changes from baseline of Number of TMPRSS2-ERG mRNA copies in blood/PBMC | Baseline to 6 months

SECONDARY OUTCOMES:
Number of Adverse Events from screening to the end of study visit (as reported by the investigator based on Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.3) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe Ltd.
Locations (3):
- Netherlands (3):
  - Site NL31005 St. Antonius ziekenhuis, Nieuwegein
  - Site NL31004 Radboudumc, Nijmegen
  - Site NL31001 Canisius-Wilhelmina Ziekenhuis, Nijmegen

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=181